CLINICAL TRIAL: NCT07387042
Title: Comparison of Laparoscopic Nissen Fundoplication and Hill-Snow Repair for Hiatus Hernia With Endoscopic Evaluation: Randomized Controlled Trial
Brief Title: Comparison of Laparoscopic Nissen Fundoplication and Hill-Snow Repair for Hiatus Hernia With Endoscopic Evaluation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Hassaan Hamdy, Assistrent Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1799/11/2025
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Hiatal Hernia With Gastroesophageal Reflux Disease
Keywords: Hiatus Hernia; Nissen Fundoplication; Hill-Snow repair; Endoscopy
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Hill-Snow repair (Experimental)
  Interventions: Procedure: Laparoscopic Hill-Snow repair
- Laparoscopic Nissen Fundoplication (Active Comparator)
  Interventions: Procedure: Laparoscopic Nissen Fundoplication

INTERVENTIONS:
Procedure: Laparoscopic Hill-Snow repair — a laparoscopic surgical operation to fix severe acid reflux (GERD) and hiatal hernias by restoring the natural anti-reflux mechanism,acting as an alternative to the more common Nissen fundoplication, It's known for firmly anchoring the stomach to reliable structures, creating a flap valve, and reducing recurrence
  What it does
  * Reduces hiatal hernia: Pulls down the stomach that has slipped into the chest.
  * Recreates valve: Re-establishes the angle of His (the valve between the esophagus and stomach).
  * Secures the junction: Sews the lower esophagus and stomach to the diaphragm and abdominal structures, preventing reflux
  How it works (basic steps)
  Dissect: Free the esophagus and pull down the herniated stomach. Repair hernia: Close the opening (hiatus) in the diaphragm (cruroplasty). Fix stomach: Sew the stomach (fundus) to the esophagus and diaphragm (gastropexy).
  Create angle: Recreate the angle of His with sutures
  Arms: Laparoscopic Hill-Snow repair
Procedure: Laparoscopic Nissen Fundoplication — a minimally invasive keyhole surgery that treats severe acid reflux (GERD) by wrapping the upper part of the stomach (fundus) around the lower esophagus to create a stronger valve, preventing stomach acid from traveling up. Performed through small incisions, it's a more permanent solution than medication, often used when lifestyle changes and drugs fail, and involves a quicker recovery than traditional open surgery.
  How it works Reinforces the valve: The stomach's fundus is wrapped around the esophagus, strengthening the natural anti-reflux barrier.
  Stops acid flow: This "wrap" stops stomach acid and enzymes from splashing back into the esophagus.
  Corrects hiatal hernia: If present, a hiatal hernia (when part of the stomach pushes through the diaphragm) is also repaired during the procedure.
  Arms: Laparoscopic Nissen Fundoplication

SUMMARY:
The goal of this clinical trial is to compare the clinical efficacy and safety of laparoscopic Nissen fundoplication (LNF) versus laparoscopic Hill-Snow repair (LHS) in the management of patients with congenital hiatus hernia, to evaluate the role of upper gastrointestinal endoscopy in the preoperative diagnosis and planning & to determine the utility of intraoperative endoscopy in guiding the surgical repair and ensuring its technical adequacy.

main questions are:

* which one of these techniques is safer with higher clinical efficacy represented by relief of GERD symptoms ?
* does upper GI endoscopy have a role in preoperative stage regarding diagnosis of condition and planning of treatment ?
* does upper GI endoscopy have a role in intraoperative stage regarding guiding the surgical repair and ensuring its adequacy ?

all participants will be randomly assigned in one of two groups:

* one group undergoing Laparoscopic Nissen Fundoplication
* the other group undergoing Laparoscopic Hill-Snow repair

each participsant will have preopertive, intraoperative and postoperative upper GI endoscopy to assess objectively clinical efficacy of both techniques and to define the integral role of endoscopy in all three perioperative stages

DETAILED DESCRIPTION:
Congenital hiatus hernia (CHH), though less common than acquired forms, presents a significant clinical challenge, particularly in the pediatric and young adult populations. It is characterized by a congenital defect in the phrenoesophageal membrane, allowing for herniation of gastric cardia into the mediastinum. This anatomical disruption compromises the lower esophageal sphincter (LES) mechanism, leading to severe gastroesophageal reflux disease (GERD), which can result in failure to thrive, esophagitis, recurrent aspiration pneumonia, and long-term sequelae like Barrett's esophagus.

When medical management fails or in cases of significant complications, surgical intervention is imperative. The goals of surgery are the anatomical reduction of the hernia, reconstruction of the esophagogastric junction (EGJ), and restoration of an effective anti-reflux barrier. Laparoscopic repair has become the gold standard due to its benefits of reduced postoperative pain, shorter hospital stay, and better cosmesis.

Two prominent laparoscopic techniques are:

Laparoscopic Nissen Fundoplication (LNF): A 360-degree wrap is the most common anti-reflux procedure worldwide. It is highly effective in controlling reflux but is associated with potential side effects like gas-bloat syndrome, dysphagia, and inability to belch.

Laparoscopic Hill-Snow Repair (LHS): This technique focuses on a precise anatomical restoration of the EGJ by anchoring it to the median arcuate ligament of the diaphragm. It aims to recreate the valvular mechanism without a complete wrap, potentially reducing the typical side effects of Nissen fundoplication.

Endoscopy plays a crucial but often under-standardized role in the perioperative management of CHH.

Preoperatively, it is essential for diagnosing esophagitis, Barrett's metaplasia, and ruling out other pathologies. It also helps in assessing the size and reducibility of the hernia.

Intraoperatively, endoscopy (laparoscopic-endoscopic collaboration) can guide the surgeon in assessing the tightness of the fundoplication, identifying the Z-line for accurate placement of the wrap, and ensuring no mucosal perforation has occurred.

Postoperatively, endoscopy is the primary tool for evaluating anatomical success, detecting recurrence, and managing persistent symptoms like dysphagia.

While numerous studies have compared various fundoplication techniques for GERD, there is a paucity of literature directly comparing LNF and LHS specifically in the context of congenital hiatus hernia. Furthermore, a systematic protocol defining the integral role of endoscopy in all three perioperative stages is lacking. This study aims to fill this gap by providing a comparative analysis of the functional outcomes and complications of these two techniques and by establishing a standardized perioperative endoscopic protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged less than 18 years including both sexes with a confirmed diagnosis of congenital hiatus hernia
* Diagnosis of hiatus hernia refractory to maximal medical therapy (PPI for ≥12 weeks) AND/OR presence of complications (e.g., erosive esophagitis, Barrett's esophagus, recurrent aspiration pneumonia, failure to thrive)
* Objective evidence of pathological GERD on upper endoscopy e.g: erosive esophagitis, Barrett's esophagus.

Exclusion Criteria:

* Previous esophageal or gastric surgery
* Contraindications to laparoscopy e.g: cardiopulmonary decompensated cases.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Degree of relief of GERD symptoms assessed by GERD Health-Related Quality Of Life (GERD-HRQL) score | 6 months postoperatively
  The GERD-HRQL questionnaire was developed and validated to measure changes of typical GERD symptoms such as heartburn and regurgitation in response to surgical or medical treatment. Total Score: Calculated by summing the individual scores to 15 questions * Greatest possible score (worst symptoms) = 75 * Lowest possible score (no symptoms) = 0 Heartburn Score: Calculated by summing the individual scores to 6 questions * Worst heartburn symptoms = 30 * No heartburn symptoms = 0 * Scores less than or equal to 12 with each individual question not exceeding 2 indicate heartburn elimination. Regurgitation Score: Calculated by summing the individual scores to 6 questions . *Worst regurgitation symptoms = 30 * No regurgitation = 0 * Scores less than or equal to 12 with each individual question not exceeding 2 indicate regurgitation.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa A El sayed, Principal Investigator — Minia University
Locations (1):
- Pediatrics and Pediatric Surgery University Hospital, Faculty Of Medicine, Minia Universty, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gyawali, C. P., Kahrilas, P. J., Savarino, E., Zerbib, F., Mion, F., Smout, A. J., ... & Sifrim, D. (2018). Modern diagnosis of GERD: the Lyon Consensus. Gut, 67(7), 1351-1362
- [Background] Mönig, S. P., & Hölscher, A. H. (2006). Intraoperative endoscopy. Langenbeck's Archives of Surgery, 391(2), 99-104.
- [Background] Spechler, S. J., & Hunter, J. G. (2017). A Modern View of Hiatal Hernia: Lessons from Surgical and Gastroenterologic Literature. Gastroenterology, 153(4), 911-914.
- [Background] Hill, L. D., & Snow, L. L. (1999). The Hill-Snow repair for gastroesophageal reflux disease. Surgical Clinics of North America.
- [Background] Nissen, R. (1956). Eine einfache Operation zur Beeinflussung der Refluxoesophagitis. Schweiz Med Wochenschr.
- [Background] Stefanidis, D., Hope, W. W., Kohn, G. P., Reardon, P. R., Richardson, W. S., & Fanelli, R. D. (2010). Guidelines for surgical treatment of gastroesophageal reflux disease. Surgical Endoscopy, 24(11), 2647-2669.
- [Background] Hyun, J. J., & Bak, Y. T. (2011). Clinical Significance of Hiatal Hernia. The Korean Journal of Gastroenterology, 57(3), 160-165.